CLINICAL TRIAL: NCT01902667
Title: Preoperative Imaging in Retroperitoneal Sarcoma
Acronym: PIRS
Status: Completed | Type: Observational
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Royal Marsden NHS Foundation Trust (Other); Cancer Research UK (Other)
Responsible Party: Principal Investigator, Nandita deSouza, Professor of Translational Imaging, Institute of Cancer Research, United Kingdom
Other Study IDs: 13/EE/0186 CCR3992
Record Dates: First submitted 2013-07-09; First posted 2013-07-18 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Cancer
Keywords: Retroperitoneal Sarcoma; Magnetic Resonance Imaging
MeSH Terms: conditions — Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Curative intent surgery alone: Patients with retroperitoneal sarcoma randomised into surgery alone arm.
  Interventions: Procedure: Magnetic Resonance Imaging
- Pre-operative radiotherapy plus surgery: Patients with retroperitoneal sarcoma randomised to Arm 2: pre-operative radiotherapy plus surgery.
  Interventions: Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Procedure: Magnetic Resonance Imaging

SUMMARY:
This is a prospective observational study in which patients with untreated retroperitoneal sarcoma will have Magnetic Resonance Imaging (MRI) prior to surgery. In addition, patients who will be undergoing pre-operative radiotherapy will have an additional MRI scan at two weeks post radiotherapy. For both groups, the magnetic resonance images will be correlated with tumour pathology.

The study hypothesis is that Magnetic Resonance Imaging will provide a more accurate assessment of tumour volume and local staging than CT and will identify areas of altered oxygenation, cellularity and perfusion which change in response to radiotherapy before tumour shrinkage occurs.

ELIGIBILITY:
Inclusion Criteria:

* Patients with retroperitoneal sarcomas planned for surgical resection +/- preoperative radiotherapy.

Exclusion Criteria:

* MRI incompatible metal implants
* claustrophobia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with retroperitoneal sarcoma randomised for preoperative radiotherapy plus surgery versus surgery alone.
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Prediction, by MRI, of early response to radiotherapy prior to tumour shrinkage | 2-4 weeks
  Changes in volume, maximum axial diameter, ADC, F, D, D*, T2, R2* and enhancing fraction from baseline to post radiotherapy will be presented. A paired T-test (or Wilcoxon Signed Rank Test) may be used to test the difference between baseline and post radiotherapy. Differences in these values will be presented for responders and non-responders, which will be tested by independent T-test. Response will be determined by tumour size, enhancing fraction and histopathological evidence of response.

SECONDARY OUTCOMES:
To determine the reproducibility of multi-parametric MRI measurements within tumour regions of interest in patients with retroperitoneal sarcoma. | 1-7 days
  Reproducibility of the parameter ADC-Apparent Diffusion Coefficient (also F, D, D*, T2 and R2* values)between the two scans at baseline (within 7 days of each other)will be assessed using the Bland Altman method.

OTHER OUTCOMES:
Correlation of imaging features with histopathological assessment of tumour size, local staging, cellularity, necrosis and viable tumour. | 2 months
  Correlation between the ADC (and D) and %ki 67 uptake, % necrosis, %fat content, % of viable tumour, % hyalinization/fibrosis, % dedifferentiated component, cellularity and stroma morphology will be assessed using the Pearson's correlation coefficient or the Spearman's (whichever is appropriate).

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom

REFERENCES:
- [Derived] Winfield JM, Miah AB, Strauss D, Thway K, Collins DJ, deSouza NM, Leach MO, Morgan VA, Giles SL, Moskovic E, Hayes A, Smith M, Zaidi SH, Henderson D, Messiou C. Utility of Multi-Parametric Quantitative Magnetic Resonance Imaging for Characterization and Radiotherapy Response Assessment in Soft-Tissue Sarcomas and Correlation With Histopathology. Front Oncol. 2019 Apr 25;9:280. doi: 10.3389/fonc.2019.00280. eCollection 2019. PMID 31106141